CLINICAL TRIAL: NCT03494725
Title: Proof-of-Concept "Stress & Anxiety Dampening Effects of Lpc-37"
Brief Title: Stress & Anxiety Dampening Effects of a Probiotic Supplement Compared to Placebo in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daacro (Network)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Principal Investigator, Juliane Hellhammer, PhD, Daacro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DU01-2017
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Healthy; Stress, Psychological
Keywords: Probiotic; Gut-brain axis; Stress; Anxiety
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lpc-37 (Active Comparator): Lacticaseibacillus paracasei Lpc-37 (Lpc-37), formerly Lactobacillus paracasei Lpc-37
  1x 1 capsule in the morning for 5 weeks
  Interventions: Dietary Supplement: Lpc-37
- Placebo (Placebo Comparator): Placebo capsule manufactured to mimic Lpc-37 capsule
  1x 1 capsule in the morning for 5 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lpc-37 — Lacticaseibacillus paracasei Lpc-37 at 1.75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide
  Arms: Lpc-37
Dietary Supplement: Placebo — microcrystalline cellulose, magnesium stearate, silicon dioxide
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether a 5 week intake of a probiotic (Lpc-37) can modulate stress and anxiety experienced by healthy subjects during and after an acute stressor compared to placebo. To measure stress and anxiety, markers of the hypothalamic-pituitary-adrenal (HPA) axis activity and questionnaires will be assessed before, during and after the Trier Social Stress Test (TSST). The results of this study indicate if the chosen study design is suitable to discover stress-related effects of probiotics.

DETAILED DESCRIPTION:
The total mass of microorganisms residing within the human intestine is approximately the same as that of the human brain. Of late, these >1000 species and >7000 strains have been described as the "brain in our belly" because of the essential role they play in physiological and psychological health and disease. The gut-brain axis describes the bidirectional communication that exists between the brain and the gut and the microbiota-gut-brain axis supports the role of the gut microbiome in this communication system. Emotional and routine daily life stress can disrupt digestive function, but increasing evidence indicates that the gut microbiota exert a profound influence on brain physiology, psychological responses and ultimately behavior.

A plethora of literature to date, albeit predominantly preclinical, have demonstrated evidence to support the role of the gut microbiome in regulating stress-related changes in physiology, behavior and brain function.

Stress is an individual process to deal with external and internal challenges that ranges from behavioral to molecular adaptations. The HPA axis and its release of stress hormones plays a major role in stress adaptation.

The purpose of this clinical trial is to determine whether a single strain of bacteria derived from the species Lacticaseibacillus paracasei Lpc-37 (Lpc-37), formerly Lactobacillus paracasei Lpc-37, can modulate stress experienced by healthy subjects exposed to the TSST measured by HPA axis activation markers and self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, written, informed consent to participate in the study
* Male or female aged between 18-45 years (inclusive)
* Body mass index (BMI) between 18.5 - 29.9 kg/m2
* Medical examination at baseline indicates they are healthy in the opinion of the investigator
* Ability of the participant (in the Principal Investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
* Agreement to comply with the protocol and study restrictions
* Available for all study visits
* Females of child-bearing potential required to provide a negative urine pregnancy test and to use contraceptives
* Easy access to internet

Exclusion Criteria:

* Self-reported diagnosis of one or more Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV axis 1 disorder(s), including but not limited to current major depression, anxiety disorder, bipolar spectrum disorder or schizophrenia
* Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal (irritable bowel syndrome (IBS), inflammatory bowel disease (IBD)), immunological, metabolic, neurodevelopmental or any condition which contraindicates, in the Investigator's judgement, entry to the study
* Currently taking (from day of screening onwards) or have previously taken (last 4 weeks prior to screening) psychoactive medication (anxiolytics, sedatives, hypnotics, anti-psychotics, anti-depressants, anti-convulsants, centrally acting corticosteroids, opioid pain relievers)
* Currently taking (from day of screening onwards) medication or dietary supplements that the Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results (e.g. melatonin, omega-3 dietary supplements, non-steroidal anti-inflammatory drugs (NSAIDS), over-the-counter (OTC) sleep medication (not categorized as sedatives, hypnotics or anti-depressants), anti-coagulants, proton pump inhibitors, anti-histamines, pseudoephedrine, cortisone, beta-blockers)
* Recent (within last 4 weeks prior to screening) or ongoing antibiotic therapy during the intervention period
* Daily consumption of concentrated sources of probiotics and/or prebiotics within 2 weeks of screening and throughout the intervention period other than the provided study products (e.g., probiotic/prebiotic tablets, capsules, drops or powders)
* Pregnant or lactating female, or pregnancy planned during intervention period
* Not fluent in German
* Have self-reported dyslexia
* History of alcohol, drug, or medication abuse
* Self-declared illicit drug users (including cannabis and cocaine) for 3 weeks prior to screening and during the intervention period
* Contraindication to any substance in the investigational product
* Hypertension (systolic ≥ 140 mmHg, diastolic ≥ 90 mmHg)
* Known hyper- or hypothyroidism unless treated and under control (stable for more than 3 months)
* Subjects having previously participated in the TSST
* Smoking > 5 cigarettes/day
* Employee of the sponsor or contract research organization (CRO)
* Participation in another study with any investigational product within 60 days of screening and during the intervention period
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study
* Participant under administrative or legal supervision

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hellhammer, PhD, Principal Investigator — Daacro GmbH & Co. KG
Locations (1):
- daacro GmbH & Co. KG, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey MT, Coe CL. Maternal separation disrupts the integrity of the intestinal microflora in infant rhesus monkeys. Dev Psychobiol. 1999 Sep;35(2):146-55. PMID 10461128
- [Background] Bailey MT, Dowd SE, Galley JD, Hufnagle AR, Allen RG, Lyte M. Exposure to a social stressor alters the structure of the intestinal microbiota: implications for stressor-induced immunomodulation. Brain Behav Immun. 2011 Mar;25(3):397-407. doi: 10.1016/j.bbi.2010.10.023. Epub 2010 Oct 30. PMID 21040780
- [Background] Bailey MT, Lubach GR, Coe CL. Prenatal stress alters bacterial colonization of the gut in infant monkeys. J Pediatr Gastroenterol Nutr. 2004 Apr;38(4):414-21. doi: 10.1097/00005176-200404000-00009. PMID 15085020
- [Background] Bercik P, Denou E, Collins J, Jackson W, Lu J, Jury J, Deng Y, Blennerhassett P, Macri J, McCoy KD, Verdu EF, Collins SM. The intestinal microbiota affect central levels of brain-derived neurotropic factor and behavior in mice. Gastroenterology. 2011 Aug;141(2):599-609, 609.e1-3. doi: 10.1053/j.gastro.2011.04.052. Epub 2011 Apr 30. PMID 21683077
- [Background] Bercik P, Park AJ, Sinclair D, Khoshdel A, Lu J, Huang X, Deng Y, Blennerhassett PA, Fahnestock M, Moine D, Berger B, Huizinga JD, Kunze W, McLean PG, Bergonzelli GE, Collins SM, Verdu EF. The anxiolytic effect of Bifidobacterium longum NCC3001 involves vagal pathways for gut-brain communication. Neurogastroenterol Motil. 2011 Dec;23(12):1132-9. doi: 10.1111/j.1365-2982.2011.01796.x. Epub 2011 Oct 11. PMID 21988661
- [Background] Bharwani A, Mian MF, Foster JA, Surette MG, Bienenstock J, Forsythe P. Structural & functional consequences of chronic psychosocial stress on the microbiome & host. Psychoneuroendocrinology. 2016 Jan;63:217-27. doi: 10.1016/j.psyneuen.2015.10.001. Epub 2015 Oct 9. PMID 26479188
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Clarke G, Grenham S, Scully P, Fitzgerald P, Moloney RD, Shanahan F, Dinan TG, Cryan JF. The microbiome-gut-brain axis during early life regulates the hippocampal serotonergic system in a sex-dependent manner. Mol Psychiatry. 2013 Jun;18(6):666-73. doi: 10.1038/mp.2012.77. Epub 2012 Jun 12. PMID 22688187
- [Background] Daulatzai MA. Chronic functional bowel syndrome enhances gut-brain axis dysfunction, neuroinflammation, cognitive impairment, and vulnerability to dementia. Neurochem Res. 2014 Apr;39(4):624-44. doi: 10.1007/s11064-014-1266-6. Epub 2014 Mar 4. PMID 24590859
- [Background] Dallman, M. F., & Hellhammer, D. (2011). Regulation of the hypothalamo-pituitaryadrenal axis, chronic stress, and energy: the role of brain networks. The handbook of stress science: Biology, psychology, and health, 11-36.
- [Background] De Vadder F, Kovatcheva-Datchary P, Goncalves D, Vinera J, Zitoun C, Duchampt A, Backhed F, Mithieux G. Microbiota-generated metabolites promote metabolic benefits via gut-brain neural circuits. Cell. 2014 Jan 16;156(1-2):84-96. doi: 10.1016/j.cell.2013.12.016. Epub 2014 Jan 9. PMID 24412651
- [Background] Desbonnet L, Garrett L, Clarke G, Bienenstock J, Dinan TG. The probiotic Bifidobacteria infantis: An assessment of potential antidepressant properties in the rat. J Psychiatr Res. 2008 Dec;43(2):164-74. doi: 10.1016/j.jpsychires.2008.03.009. Epub 2008 May 5. PMID 18456279
- [Background] Desbonnet L, Garrett L, Clarke G, Kiely B, Cryan JF, Dinan TG. Effects of the probiotic Bifidobacterium infantis in the maternal separation model of depression. Neuroscience. 2010 Nov 10;170(4):1179-88. doi: 10.1016/j.neuroscience.2010.08.005. Epub 2010 Aug 6. PMID 20696216
- [Background] Dickerson SS, Kemeny ME. Acute stressors and cortisol responses: a theoretical integration and synthesis of laboratory research. Psychol Bull. 2004 May;130(3):355-91. doi: 10.1037/0033-2909.130.3.355. PMID 15122924
- [Background] Dinan TG, Cryan JF. Mood by microbe: towards clinical translation. Genome Med. 2016 Apr 6;8(1):36. doi: 10.1186/s13073-016-0292-1. PMID 27048547
- [Background] Dinan TG, Stanton C, Cryan JF. Psychobiotics: a novel class of psychotropic. Biol Psychiatry. 2013 Nov 15;74(10):720-6. doi: 10.1016/j.biopsych.2013.05.001. Epub 2013 Jun 10. PMID 23759244
- [Background] Dinan TG, Stilling RM, Stanton C, Cryan JF. Collective unconscious: how gut microbes shape human behavior. J Psychiatr Res. 2015 Apr;63:1-9. doi: 10.1016/j.jpsychires.2015.02.021. Epub 2015 Mar 3. PMID 25772005
- [Background] Foster JA, Lyte M, Meyer E, Cryan JF. Gut Microbiota and Brain Function: An Evolving Field in Neuroscience. Int J Neuropsychopharmacol. 2016 Apr 29;19(5):pyv114. doi: 10.1093/ijnp/pyv114. Print 2016 May. PMID 26438800
- [Background] Foster JA, McVey Neufeld KA. Gut-brain axis: how the microbiome influences anxiety and depression. Trends Neurosci. 2013 May;36(5):305-12. doi: 10.1016/j.tins.2013.01.005. Epub 2013 Feb 4. PMID 23384445
- [Background] Foster JA, Rinaman L, Cryan JF. Stress & the gut-brain axis: Regulation by the microbiome. Neurobiol Stress. 2017 Mar 19;7:124-136. doi: 10.1016/j.ynstr.2017.03.001. eCollection 2017 Dec. PMID 29276734
- [Background] Fries E, Dettenborn L, Kirschbaum C. The cortisol awakening response (CAR): facts and future directions. Int J Psychophysiol. 2009 Apr;72(1):67-73. doi: 10.1016/j.ijpsycho.2008.03.014. Epub 2008 Sep 30. PMID 18854200
- [Background] Golubeva AV, Crampton S, Desbonnet L, Edge D, O'Sullivan O, Lomasney KW, Zhdanov AV, Crispie F, Moloney RD, Borre YE, Cotter PD, Hyland NP, O'Halloran KD, Dinan TG, O'Keeffe GW, Cryan JF. Prenatal stress-induced alterations in major physiological systems correlate with gut microbiota composition in adulthood. Psychoneuroendocrinology. 2015 Oct;60:58-74. doi: 10.1016/j.psyneuen.2015.06.002. Epub 2015 Jun 17. PMID 26135201
- [Background] Diaz Heijtz R, Wang S, Anuar F, Qian Y, Bjorkholm B, Samuelsson A, Hibberd ML, Forssberg H, Pettersson S. Normal gut microbiota modulates brain development and behavior. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3047-52. doi: 10.1073/pnas.1010529108. Epub 2011 Jan 31. PMID 21282636
- [Background] Hellhammer DH, Wade S. Endocrine correlates of stress vulnerability. Psychother Psychosom. 1993;60(1):8-17. doi: 10.1159/000288675. PMID 8234641
- [Background] Holsboer F, Ising M. Stress hormone regulation: biological role and translation into therapy. Annu Rev Psychol. 2010;61:81-109, C1-11. doi: 10.1146/annurev.psych.093008.100321. PMID 19575614
- [Background] Janak PH, Tye KM. From circuits to behaviour in the amygdala. Nature. 2015 Jan 15;517(7534):284-92. doi: 10.1038/nature14188. PMID 25592533
- [Background] Jasarevic E, Howerton CL, Howard CD, Bale TL. Alterations in the Vaginal Microbiome by Maternal Stress Are Associated With Metabolic Reprogramming of the Offspring Gut and Brain. Endocrinology. 2015 Sep;156(9):3265-76. doi: 10.1210/en.2015-1177. Epub 2015 Jun 16. PMID 26079804
- [Background] Kelly JR, Borre Y, O' Brien C, Patterson E, El Aidy S, Deane J, Kennedy PJ, Beers S, Scott K, Moloney G, Hoban AE, Scott L, Fitzgerald P, Ross P, Stanton C, Clarke G, Cryan JF, Dinan TG. Transferring the blues: Depression-associated gut microbiota induces neurobehavioural changes in the rat. J Psychiatr Res. 2016 Nov;82:109-18. doi: 10.1016/j.jpsychires.2016.07.019. Epub 2016 Jul 25. PMID 27491067
- [Background] Kelly JR, Kennedy PJ, Cryan JF, Dinan TG, Clarke G, Hyland NP. Breaking down the barriers: the gut microbiome, intestinal permeability and stress-related psychiatric disorders. Front Cell Neurosci. 2015 Oct 14;9:392. doi: 10.3389/fncel.2015.00392. eCollection 2015. PMID 26528128
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Kudielka BM, Wust S. Human models in acute and chronic stress: assessing determinants of individual hypothalamus-pituitary-adrenal axis activity and reactivity. Stress. 2010 Jan;13(1):1-14. doi: 10.3109/10253890902874913. PMID 20105052
- [Background] Luczynski P, McVey Neufeld KA, Oriach CS, Clarke G, Dinan TG, Cryan JF. Growing up in a Bubble: Using Germ-Free Animals to Assess the Influence of the Gut Microbiota on Brain and Behavior. Int J Neuropsychopharmacol. 2016 Aug 12;19(8):pyw020. doi: 10.1093/ijnp/pyw020. Print 2016 Aug. PMID 26912607
- [Background] Mackowiak PA. Recycling metchnikoff: probiotics, the intestinal microbiome and the quest for long life. Front Public Health. 2013 Nov 13;1:52. doi: 10.3389/fpubh.2013.00052. PMID 24350221
- [Background] Marcos A, Warnberg J, Nova E, Gomez S, Alvarez A, Alvarez R, Mateos JA, Cobo JM. The effect of milk fermented by yogurt cultures plus Lactobacillus casei DN-114001 on the immune response of subjects under academic examination stress. Eur J Nutr. 2004 Dec;43(6):381-9. doi: 10.1007/s00394-004-0517-8. Epub 2004 Jul 14. PMID 15309418
- [Background] Marin IA, Goertz JE, Ren T, Rich SS, Onengut-Gumuscu S, Farber E, Wu M, Overall CC, Kipnis J, Gaultier A. Microbiota alteration is associated with the development of stress-induced despair behavior. Sci Rep. 2017 Mar 7;7:43859. doi: 10.1038/srep43859. PMID 28266612
- [Background] Mason JW. A review of psychoendocrine research on the pituitary-adrenal cortical system. Psychosom Med. 1968 Sep-Oct;30(5):Suppl:576-607. No abstract available. PMID 4303377
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Nater UM, La Marca R, Florin L, Moses A, Langhans W, Koller MM, Ehlert U. Stress-induced changes in human salivary alpha-amylase activity -- associations with adrenergic activity. Psychoneuroendocrinology. 2006 Jan;31(1):49-58. doi: 10.1016/j.psyneuen.2005.05.010. Epub 2005 Jul 5. PMID 16002223
- [Background] Neufeld KM, Kang N, Bienenstock J, Foster JA. Reduced anxiety-like behavior and central neurochemical change in germ-free mice. Neurogastroenterol Motil. 2011 Mar;23(3):255-64, e119. doi: 10.1111/j.1365-2982.2010.01620.x. Epub 2010 Nov 5. PMID 21054680
- [Background] Nishida, K., Sawada, D., Kuwano, Y., Tanaka, H., Sugawara, T., Aoki, Y., ... & Rokutan, K. (2017). Daily administration of paraprobiotic lactobacillus gasseri cp2305 ameliorates chronic stress-associated symptoms in Japanese medical students. Journal of Functional Foods, 36, 112-121.
- [Background] O'Mahony SM, Marchesi JR, Scully P, Codling C, Ceolho AM, Quigley EM, Cryan JF, Dinan TG. Early life stress alters behavior, immunity, and microbiota in rats: implications for irritable bowel syndrome and psychiatric illnesses. Biol Psychiatry. 2009 Feb 1;65(3):263-7. doi: 10.1016/j.biopsych.2008.06.026. Epub 2008 Aug 23. PMID 18723164
- [Background] O'Mahony SM, Clarke G, Borre YE, Dinan TG, Cryan JF. Serotonin, tryptophan metabolism and the brain-gut-microbiome axis. Behav Brain Res. 2015 Jan 15;277:32-48. doi: 10.1016/j.bbr.2014.07.027. Epub 2014 Jul 29. PMID 25078296
- [Background] Ogbonnaya ES, Clarke G, Shanahan F, Dinan TG, Cryan JF, O'Leary OF. Adult Hippocampal Neurogenesis Is Regulated by the Microbiome. Biol Psychiatry. 2015 Aug 15;78(4):e7-9. doi: 10.1016/j.biopsych.2014.12.023. Epub 2015 Jan 9. No abstract available. PMID 25700599
- [Background] De Palma G, Collins SM, Bercik P, Verdu EF. The microbiota-gut-brain axis in gastrointestinal disorders: stressed bugs, stressed brain or both? J Physiol. 2014 Jul 15;592(14):2989-97. doi: 10.1113/jphysiol.2014.273995. Epub 2014 Apr 22. PMID 24756641
- [Background] Pinto-Sanchez MI, Hall GB, Ghajar K, Nardelli A, Bolino C, Lau JT, Martin FP, Cominetti O, Welsh C, Rieder A, Traynor J, Gregory C, De Palma G, Pigrau M, Ford AC, Macri J, Berger B, Bergonzelli G, Surette MG, Collins SM, Moayyedi P, Bercik P. Probiotic Bifidobacterium longum NCC3001 Reduces Depression Scores and Alters Brain Activity: A Pilot Study in Patients With Irritable Bowel Syndrome. Gastroenterology. 2017 Aug;153(2):448-459.e8. doi: 10.1053/j.gastro.2017.05.003. Epub 2017 May 5. PMID 28483500
- [Background] Sherwin E, Rea K, Dinan TG, Cryan JF. A gut (microbiome) feeling about the brain. Curr Opin Gastroenterol. 2016 Mar;32(2):96-102. doi: 10.1097/MOG.0000000000000244. PMID 26760398
- [Background] Sherwin E, Sandhu KV, Dinan TG, Cryan JF. May the Force Be With You: The Light and Dark Sides of the Microbiota-Gut-Brain Axis in Neuropsychiatry. CNS Drugs. 2016 Nov;30(11):1019-1041. doi: 10.1007/s40263-016-0370-3. PMID 27417321
- [Background] Slykerman RF, Hood F, Wickens K, Thompson JMD, Barthow C, Murphy R, Kang J, Rowden J, Stone P, Crane J, Stanley T, Abels P, Purdie G, Maude R, Mitchell EA; Probiotic in Pregnancy Study Group. Effect of Lactobacillus rhamnosus HN001 in Pregnancy on Postpartum Symptoms of Depression and Anxiety: A Randomised Double-blind Placebo-controlled Trial. EBioMedicine. 2017 Oct;24:159-165. doi: 10.1016/j.ebiom.2017.09.013. Epub 2017 Sep 14. PMID 28943228
- [Background] Steenbergen L, Sellaro R, van Hemert S, Bosch JA, Colzato LS. A randomized controlled trial to test the effect of multispecies probiotics on cognitive reactivity to sad mood. Brain Behav Immun. 2015 Aug;48:258-64. doi: 10.1016/j.bbi.2015.04.003. Epub 2015 Apr 7. PMID 25862297
- [Background] Stilling RM, Ryan FJ, Hoban AE, Shanahan F, Clarke G, Claesson MJ, Dinan TG, Cryan JF. Microbes & neurodevelopment--Absence of microbiota during early life increases activity-related transcriptional pathways in the amygdala. Brain Behav Immun. 2015 Nov;50:209-220. doi: 10.1016/j.bbi.2015.07.009. Epub 2015 Jul 14. PMID 26184083
- [Background] Sudo N, Chida Y, Aiba Y, Sonoda J, Oyama N, Yu XN, Kubo C, Koga Y. Postnatal microbial colonization programs the hypothalamic-pituitary-adrenal system for stress response in mice. J Physiol. 2004 Jul 1;558(Pt 1):263-75. doi: 10.1113/jphysiol.2004.063388. Epub 2004 May 7. PMID 15133062
- [Background] Takada M, Nishida K, Kataoka-Kato A, Gondo Y, Ishikawa H, Suda K, Kawai M, Hoshi R, Watanabe O, Igarashi T, Kuwano Y, Miyazaki K, Rokutan K. Probiotic Lactobacillus casei strain Shirota relieves stress-associated symptoms by modulating the gut-brain interaction in human and animal models. Neurogastroenterol Motil. 2016 Jul;28(7):1027-36. doi: 10.1111/nmo.12804. Epub 2016 Feb 20. PMID 26896291
- [Background] Takai N, Yamaguchi M, Aragaki T, Eto K, Uchihashi K, Nishikawa Y. Effect of psychological stress on the salivary cortisol and amylase levels in healthy young adults. Arch Oral Biol. 2004 Dec;49(12):963-8. doi: 10.1016/j.archoralbio.2004.06.007. PMID 15485637
- [Background] Tannock GW, Savage DC. Influences of dietary and environmental stress on microbial populations in the murine gastrointestinal tract. Infect Immun. 1974 Mar;9(3):591-8. doi: 10.1128/iai.9.3.591-598.1974. PMID 4593471
- [Background] Tillisch K, Labus J, Kilpatrick L, Jiang Z, Stains J, Ebrat B, Guyonnet D, Legrain-Raspaud S, Trotin B, Naliboff B, Mayer EA. Consumption of fermented milk product with probiotic modulates brain activity. Gastroenterology. 2013 Jun;144(7):1394-401, 1401.e1-4. doi: 10.1053/j.gastro.2013.02.043. Epub 2013 Mar 6. PMID 23474283
- [Background] Tsigos C, Chrousos GP. Hypothalamic-pituitary-adrenal axis, neuroendocrine factors and stress. J Psychosom Res. 2002 Oct;53(4):865-71. doi: 10.1016/s0022-3999(02)00429-4. PMID 12377295
- [Derived] Patterson E, Griffin SM, Ibarra A, Ellsiepen E, Hellhammer J. Lacticaseibacillus paracasei Lpc-37(R) improves psychological and physiological markers of stress and anxiety in healthy adults: a randomized, double-blind, placebo-controlled and parallel clinical trial (the Sisu study). Neurobiol Stress. 2020 Nov 24;13:100277. doi: 10.1016/j.ynstr.2020.100277. eCollection 2020 Nov. PMID 33385020
- See also: daacro homepage — http://www.daacro.de

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 176 eligible participants, 120 met inclusion criteria and were enrolled in the study between April and October 2018.
Groups:
- Lpc-37: Verum: Lacticaseibacillus paracasei Lpc-37
  Ingredients: Lacticaseibacillus paracasei Lpc-37 at 1,75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide
  Participants took one capsule of the Investigational Product (IP) every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified for both groups by gender and underlying chronic stress, as assessed using the Trier Inventory for Chronic Stress (TICS).
- Placebo: Placebo: capsule manufactured to mimic Lpc-37 capsule
  Ingredients: microcrystalline cellulose, magnesium stearate, silicon dioxide
  Participants took one capsule of the Investigational Product (IP) every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified for both groups by gender and underlying chronic stress, as assessed using the Trier Inventory for Chronic Stress (TICS).
Period: Overall Study
Arm/Group | Lpc-37 | Placebo
Started | 60 | 60
Intervention (Post 2 Weeks run-in) (N=2 did not receive any treatment. Reasons: antibiotic therapy and consent withdrawn during run-in.) | 59 | 59
Completed | 59 | 58
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Antibiotic use | 1 | 0

BASELINE CHARACTERISTICS:
Population: 120 participants met the inclusion/exlusion criteria and were enrolled in the study. Two participants were excluded during the run-in period (use of antibiotics and withdrawn consent) and one participant withdrew consent during the intervention period.
Groups:
- Lpc-37: Verum: Lacticaseibacillus paracasei Lpc-37 (Lpc-37)
  Ingredients: Lacticaseibacillus paracasei Lpc-37 at 1,75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide
  Participants took one capsule of the IP every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified for both groups by gender and underlying chronic stress, as assessed using the Trier Inventory for Chronic Stress (TICS).
- Placebo: Placebo: capsule manufactured to mimic Lpc-37 capsule
  Ingredients: microcrystalline cellulose, magnesium stearate, silicon dioxide
  Participants took one capsule of the IP every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified for both groups by gender and underlying chronic stress, as assessed using the Trier Inventory for Chronic Stress (TICS).
- Total: Total of all reporting groups
Arm/Group | Lpc-37 | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.73 (4.27) | 23.25 (4.20) | 23.49 (4.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 30 | 30 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 60 | 60 | 120
Weight [Mean (Standard Deviation); unit: kg] | 71.13 (11.05) | 69.79 (12.15) | 70.46 (11.58)
Height [Mean (Standard Deviation); unit: cm] | 175.58 (8.86) | 173.58 (9.33) | 174.58 (9.11)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 22.97 (2.30) | 23.02 (2.67) | 23.00 (2.48)
Systolic blood pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 120.75 (12.09) | 120.72 (13.47) | 120.73 (12.74)
Diastolic blood pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 74.22 (7.25) | 74.88 (8.53) | 74.55 (7.88)
Heart rate [Mean (Standard Deviation); unit: bpm] | 72.27 (13.71) | 71.03 (12.43) | 71.65 (13.05)

OUTCOME MEASURES:

1. Primary Outcome: Change of the Heart Rate (HR) in Response to the Trier Social Stress Test (TSST)
Description: Efficacy was defined as a lower increase in HR in response to the TSST following intervention with Lpc-37, compared to placebo.
Time Frame: Continuous measurement starting 20 minutes before and ending 20 minutes after the TSST after 5 weeks of product intake. Mean values were calculated per group at seven-time windows before, during and after the TSST
Population: PerProtocol population included all randomized participants that satisfied inclusion/exclusion criteria and had no major protocol deviations (total 113; Lpc-37 n=55; placebo n=58). For individual endpoints, participants were excluded if they showed deviations that were considered to possibly affect the endpoint in question (number analyzed varies).
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Lpc-37: Verum: Lacticaseibacillus paracasei Lpc-37 Ingredients: Lacticaseibacillus paracasei Lpc-37 at 1,75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide Participants took one capsule of the IP every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified for both groups by gender and underlying chronic stress, as assessed using the Trier Inventory for Chronic Stress (TICS).
- Placebo: Placebo: capsule manufactured to mimic Lpc-37 capsule
  Ingredients: microcrystalline cellulose, magnesium stearate, silicon dioxide
  Participants took one capsule of the IP every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified by gender and stress level to both groups.
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 57
bpm
  Pre-TSST -20min | 74.84 (10.20) | 74.34 (9.04)
  Pre-TSST -10min | 88.15 (11.13) | 86.69 (10.74)
  Pre-TSST -3min | 97.34 (17.15) | 97.62 (16.23)
  during TSST (Interview) | 107.56 (21.56) | 105.66 (18.86)
  during TSST (Arithmetic) | 102.77 (19.57) | 100.81 (17.20)
  Post-TSST +10min | 93.32 (14.08) | 90.81 (12.11)
  Post-TSST +20min | 75.88 (11.11) | 74.97 (9.86)
Statistical Analysis 1: Comparison: Lpc-37 vs Placebo; The sample size was computed for a repeated measurement ANOVA with two groups and seven repeated measurements (power=0.85, α=0.05, f=0.1). The calculation resulted in a group size of 56 participants each, which was rounded up to 60 participants per treatment group to account for attrition; Test type: Superiority; p = 0.757, Mixed Models Analysis — Outcome was subjected to transformation to meet model assumptions. The threshold for statistical significance was p=0.05; Linear mixed model

2. Secondary Outcome: Changes in Pre and Post Treatment STAI-state Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of State-Trait-Anxiety-Inventory (STAI)-state scores compared to placebo.
  Measured with the german version of the State-Trait-Anxiety Inventory, scale anxiety as a temporary emotional state (STAI-X1). Answers are given on a four-point rating scale ranging from 1="not at all" to 4="very true". The score range is 20-80; Higher scores indicate more anxiety.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Groups:
- Lpc-37: Verum: Lacticaseibacillus paracasei Lpc-37
  Ingredients: Lacticaseibacillus paracasei Lpc-37 at 1,75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide
  Participants took one capsule of the IP every morning for 5 weeks, 30 minutes before breakfast or their first meal of the day, with a glass of plain (non-sparkling) water.
  Participants were stratified by gender and stress level to both groups.
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 33.65 (6.80) | 34.33 (7.73)
  End of Study | 35.18 (8.38) | 35.33 (8.37)

3. Secondary Outcome: Changes in Pre and Post Treatment Perceived Stress Scale (PSS) Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of Perceived Stress Scale (PSS) scores compared to placebo.
  Measured with the german version of the PSS as a psychological instrument for measuring stress perception. It assesses how unpredictable, uncontrollable and overloaded participants perceived their lives to have been within the last month. The PSS comprises 14 items that are answered on a five-point rating scale ranging from 0 = "never" to 4 = "very often". Individual scores on the PSS can range from 0 to 56 with higher scores indicating higher perceived stress.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 57
score
  Baseline | 21.89 (7.90) | 20.72 (7.97)
  End of Study | 20.49 (7.51) | 21.56 (8.16)

4. Secondary Outcome: Changes in Pre and Post Treatment DASS Depression Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of Depression Anxiety Stress Scale (DASS) depression scores compared to placebo.
  Measured with the german version of the DASS as a 42-item self report instrument designed to measure negative emotional states of depression, anxiety and stress during the past week. The DASS includes three scales (depression, anxiety and stress) of which each scale includes 14 items that are divided into subscales of 2-5 items of similar content.
  Items are answered on a four point rating scale ranging from 0 = "not at all" to 3 = "very much". Scores of each scale are calculated by summing the scores for the relevant items.
  The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia. The items are 3, 5, 10, 13, 16, 17, 21, 24, 26, 31, 34, 37, 38, 42 and individual scores can range from 0 to 42 with higher scores indicating greater severity of the symptoms.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 4.60 (4.94) | 5.21 (6.38)
  End of Study | 4.15 (5.52) | 5.10 (5.61)

5. Secondary Outcome: Changes in Pre and Post Treatment DASS Anxiety Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of Depression Anxiety Stress Scale (DASS) anxiety scores compared to placebo.
  Measured with the german version of the DASS as a 42-item self report instrument designed to measure negative emotional states of depression, anxiety and stress during the past week. The DASS includes three scales (depression, anxiety and stress) of which each scale includes 14 items that are divided into subscales of 2-5 items of similar content.
  Items are answered on a four point rating scale ranging from 0 = "not at all" to 3 = "very much". Scores of each scale are calculated by summing the scores for the relevant items.
  The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The items are 2, 4, 7, 9, 15, 19, 20, 23, 25, 28, 30, 36, 40, 41 and individual scores can range from 0 to 42 with higher scores indicating greater severity of the symptoms.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 2.60 (3.35) | 3.07 (4.58)
  End of Study | 2.44 (3.59) | 3.45 (5.08)

6. Secondary Outcome: Changes in Pre and Post Treatment DASS Stress Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of Depression Anxiety Stress Scale (DASS) stress scores compared to placebo.
  Measured with the german version of the DASS as a 42-item self report instrument designed to measure negative emotional states of depression, anxiety and stress during the past week. The DASS includes three scales (depression, anxiety and stress) of which each scale includes 14 items that are divided into subscales of 2-5 items of similar content.
  Items are answered on a four point rating scale ranging from 0 = "not at all" to 3 = "very much". Scores of each scale are calculated by summing the scores for the relevant items.
  The stress scale (items) is sensitive to levels of chronic non-specific arousal.The stress scale items are 1, 6, 8, 11, 12, 14, 18, 22, 27, 29, 32, 33, 35, 39 and individual scores can range from 0 to 42 with higher scores indicating greater severity of the symptoms.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 9.76 (7.92) | 9.41 (7.87)
  End of Study | 8.91 (7.14) | 10.09 (8.17)

7. Secondary Outcome: Changes in Pre and Post Treatment BAI Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of Beck Anxiety Inventory (BAI) scores compared to placebo.
  Measured with the german version of the Beck Anxiety Inventory as a self-rating scale designed to measure anxiety. It comprises 21 sentences describing feelings that can occur when being anxious. These sentences are rated on a four-point rating scale ranging from 0="not at all" to 3="severely", considering the last 7 days. The score range is 0-63; Higher scores indicate higher anxiety.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 5.51 (4.46) | 5.85 (5.73)
  End of Study | 4.75 (4.39) | 6.33 (7.26)

8. Secondary Outcome: Changes in Pre and Post Treatment VAS Stress Perception Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of Visual Analog Scale (VAS) stress perception scores compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating higher perceived stress.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 19.11 (22.97) | 19.34 (21.44)
  End of Study | 23.32 (23.18) | 20.67 (21.63)

9. Secondary Outcome: Changes in Pre and Post Treatment VAS Anxiety Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of VAS anxiety scores compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating greater anxiety.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 7.29 (15.13) | 7.58 (14.05)
  End of Study | 9.26 (16.48) | 7.85 (13.40)

10. Secondary Outcome: Changes in Pre and Post Treatment VAS Insecurity Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of VAS insecurity scores compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating greater insecurity.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 13.58 (21.41) | 15.91 (19.60)
  End of Study | 16.44 (19.67) | 17.30 (20.15)

11. Secondary Outcome: Changes in Pre and Post Treatment VAS Exhaustion Scores
Description: Efficacy of the intake of Lpc-37 on the reduction of VAS exhaustion scores compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating greater exhaustion.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Baseline | 29.56 (27.63) | 23.19 (21.08)
  End of Study | 24.66 (22.78) | 18.45 (21.31)

12. Secondary Outcome: Changes in Pre and Post Treatment Systolic BP
Description: Efficacy of the intake of Lpc-37 on the reduction of systolic blood pressure (BP).
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
mmHg
  Baseline | 119.60 (14.21) | 119.66 (13.82)
  End of Study | 121.87 (14.28) | 122.86 (14.14)

13. Secondary Outcome: Changes in Pre and Post Treatment Diastolic BP
Description: Efficacy of the intake of Lpc-37 on the reduction of diastolic BP.
Time Frame: Before and after 5 weeks of study product intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
mmHg
  Baseline | 71.89 (7.74) | 71.68 (9.16)
  End of Study | 73.18 (7.45) | 74.62 (6.39)

14. Secondary Outcome: Change of STAI-State Scores in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of STAI-State scores in response to the TSST compared to placebo.
  Measured with the german version of the State-Trait-Anxiety Inventory, scale anxiety as a temporary emotional state (STAI-X1). Answers are given on a four-point rating scale ranging from 1="not at all" to 4="very true". The score range is 20-80; Higher scores indicate more anxiety.
Time Frame: 10 minutes before the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Pre-TSST -10min | 36.09 (8.45) | 36.83 (9.48)
  Post-TSST +1min | 42.38 (10.91) | 43.60 (10.00)

15. Secondary Outcome: Change of Systolic BP in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of the systolic BP in response to the TSST compared to placebo.
Time Frame: 3 minutes before the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Lpc-37: Lactobacillus paracasei Lpc-37
  1x 1 capsule in the morning for 5 weeks
  Lpc-37: Lactobacillus paracasei Lpc-37 at 1.75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide
- Placebo: Placebo capsule manufactured to mimic Lpc-37 capsule
  1x 1 capsule in the morning for 5 weeks
  Placebo: microcrystalline cellulose, magnesium stearate, silicon dioxide
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
mmHg
  Pre-TSST -3min | 115.11 (12.53) | 114.33 (14.07)
  Post-TSST +1min | 127.47 (13.67) | 129.19 (14.33)

16. Secondary Outcome: Change of Diastolic Blood Pressure (BP) in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of the diastolic BP in response to the TSST compared to placebo.
Time Frame: 3 minutes before the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Lpc-37: Lacticaseibacillus paracasei Lpc-37 (Lpc-37), formerly Lactobacillus paracasei Lpc-37
  1x 1 capsule in the morning for 5 weeks
  Lpc-37: Lacticaseibacillus paracasei Lpc-37 at 1.75 x 10^10 colony forming units (CFU) per day, microcrystalline cellulose, magnesium stearate, silicon dioxide
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
mmHg
  Pre-TSST -3min | 79.13 (7.83) | 78.41 (8.32)
  Post-TSST +1min | 90.38 (7.17) | 88.36 (9.72)

17. Secondary Outcome: Change of VAS Stress Perception Scores in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of VAS Stress perception scores in response to the TSST compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating higher perceived stress.
Time Frame: 10 minutes before the TSST, during the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Pre-TSST -10min | 19.89 (20.61) | 18.52 (21.73)
  Interview TSST (during) | 47.71 (27.08) | 51.51 (28.10)
  Post-TSST +1min | 31.72 (24.25) | 32.85 (23.66)

18. Secondary Outcome: Change of VAS Anxiety Scores in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of VAS anxiety scores in response to the TSST compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating greater anxiety.
Time Frame: 10 minutes before the TSST, during the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Pre-TSST -10min | 6.80 (10.95) | 8.50 (14.94)
  Interview TSST (during) | 20.85 (23.61) | 22.47 (23.51)
  Post-TSST +1min | 10.68 (15.19) | 11.74 (18.46)

19. Secondary Outcome: Change of VAS Insecurity Scores in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of VAS insecurity scores in response to the TSST compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating greater insecurity.
Time Frame: 10 minutes before the TSST, during the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Pre-TSST -10min | 14.47 (16.96) | 17.19 (21.37)
  Interview TSST (during) | 45.08 (28.92) | 52.19 (27.16)
  Post-TSST +1min | 23.92 (23.87) | 23.69 (23.58)

20. Secondary Outcome: Change of VAS Exhaustion Scores in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of VAS exhaustion scores in response to the TSST compared to placebo.
  Measured with a german version of the Visual Analog Scale (VAS) as a 10cm bipolar scale ranging from "not at all" to "highly". The participant indicated his/her actual perception by placing a mark on a line. VAS scores were obtained by using a ruler and measuring the position of the participants's mark with millimeter precision. To control for possible variations due to printing, the total length of the line was also measured and percentage scores for each participant were computed. Percentage scores range from 0-100. Higher scores indicating greater exhaustion.
Time Frame: 10 minutes before the TSST, during the TSST and 1 minute after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 58
score
  Pre-TSST -10min | 21.18 (21.49) | 19.79 (21.88)
  Interview TSST (during) | 19.20 (21.11) | 21.30 (22.47)
  Post-TSST +1min | 22.12 (22.46) | 25.68 (26.07)

21. Secondary Outcome: Change of Salivary Cortisol in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of salivary cortisol in response to the TSST compared to placebo.
Time Frame: 1 minute before the TSST and 1, 10, 20, 30 and 45 minutes after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 57
nmol/L
  Pre-TSST -2min | 4.79 (2.62) | 4.82 (2.60)
  Post-TSST +1min | 6.96 (3.73) | 6.85 (3.50)
  Post-TSST +10min | 9.48 (5.75) | 8.97 (5.84)
  Post-TSST +20min | 9.89 (6.51) | 9.21 (6.59)
  Post-TSST +30min | 8.04 (5.36) | 7.71 (5.06)
  Post-TSST +45min | 6.21 (3.17) | 6.16 (3.79)

22. Secondary Outcome: Change of sAA in Response to the TSST
Description: Efficacy of the intake of Lpc-37 on reduction of the increase of salivary Alpha-Amylase (sAA) in response to the TSST compared to placebo.
Time Frame: 1 minute before the TSST and 1, 10, 20, 30 and 45 minutes after the TSST after 5 weeks of study product intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 55 | 57
U/ml
  Pre-TSST -2min | 154.04 (98.17) | 161.67 (110.89)
  Post-TSST +1min | 246.29 (153.62) | 270.55 (174.85)
  Post-TSST +10min | 146.53 (86.80) | 158.85 (91.21)
  Post-TSST +20min | 130.11 (82.45) | 141.49 (93.00)
  Post-TSST +30min | 125.19 (79.67) | 138.48 (90.31)
  Post-TSST +45min | 141.13 (92.94) | 148.15 (105.60)

23. Secondary Outcome: Change of Sleep Duration Over the Course of the Treatment
Description: Efficacy of the intake of Lpc-37 on the increase of sleep duration over the course of the treatment.
  Sleep duration was monitored through the wash-out phase (week 1 and 2) and the subsequent treatment phase (weeks 3-7). Efficacy is defined as an increase, or (in case of a general decrease) reduced decrease for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group. Time is coded as a continuous variable with one value for each day and participant. Summary measures for Sleep duration for the averaged ratings per participant and week
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
min
  Week 1 (run-in) | 447.27 (47.50) | 447.45 (38.76)
  Week 2 (run-in) | 444.01 (44.60) | 448.13 (41.62)
  Week 3 (treatment) | 449.45 (41.47) | 456.90 (37.08)
  Week 4 (treatment) | 450.62 (36.07) | 459.81 (39.44)
  Week 5 (treatment) | 454.50 (39.82) | 457.26 (42.04)
  Week 6 (treatment) | 450.88 (38.95) | 450.16 (42.04)
  Week 7 (treatment) | 445.60 (40.02) | 459.66 (39.71)

24. Secondary Outcome: Change of Sleep Related Recovery Scores Over the Course of the Treatment
Description: Efficacy of the intake of Lpc-37 on the increase of sleep related recovery scores over the course of the treatment.
  Measured with a daily online diary. Sleep related recovery was rated by participants on an 11-point scale (0-10; "not at all" to "very") and monitored throughout the wash-out phase (Week 1 and 2) and the subsequent treatment phase (weeks 3-7). High scores indicate a high recovery.
  Efficacy is defined as an increase, or (in case of a general decrease) reduced decrease for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group. Time is coded as a continuous variable with one value for each day and participant. Summary measures for sleep related recovery for the averaged ratings per participant and week.
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
score
  Week 1 (run-in) | 6.71 (1.34) | 6.91 (1.00)
  Week 2 (run-in) | 7.07 (1.28) | 7.15 (1.07)
  Week 3 (treatment) | 7.32 (1.11) | 7.27 (1.12)
  Week 4 (treatment) | 7.30 (1.30) | 7.29 (1.18)
  Week 5 (treatment) | 7.36 (1.22) | 7.36 (1.19)
  Week 6 (treatment) | 7.42 (1.19) | 7.10 (1.28)
  Week 7 (treatment) | 7.31 (1.25) | 7.28 (1.18)

25. Secondary Outcome: Change of Reported Sleep Disruptions Over the Course of the Treatment by Week (Proportion Yes/Total)
Description: Efficacy of the intake of Lpc-37 on the decrease of sleep disruptions over the course of the treatment measured with a daily online diary (Proportion (yes/total)).
  Sleep disruptions were monitored through the wash-out phase and the subsequent treatment phase for each week. In the binary version, the value is either Yes or No for each day and each participant.
  Efficacy is defined as a decrease, or (in case of a general increase) reduced increase for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group. Time is coded as a continuous variable with one value for each day and participant.
  The proportion of participants with at least one sleep disruption by treatment group is given, treatment commenced after week 2. Data listed here reflect the proportion of participants who answered "Yes" (e.g. 0,477 * 44 = 20.99 participants answered with "Yes" in week 1 in the Lpc-37 group).
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: PerProtocol population included all randomized participants that satisfied inclusion/exclusion criteria and had no major protocol deviations (total 113; Lpc-37 n=55; placebo n=58). For individual endpoints, participants were excluded if they showed deviations that were considered to possibly affect the endpoint in question (number analyzed varies and is listet for each endpoint).
Measure: Number; unit: Proportion of participants (yes/total)
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
Proportion of participants (yes/total)
  Week 1 (run-in) | 0.477 | 0.465
  Week 2 (run-in) | 0.435 | 0.426
  Week 3 (treatment) | 0.354 | 0.418
  Week 4 (treatment) | 0.367 | 0.310
  Week 5 (treatment) | 0.306 | 0.292
  Week 6 (treatment) | 0.279 | 0.331
  Week 7 (treatment) | 0.290 | 0.389

26. Secondary Outcome: Change of Reported Number of Sleep Disruptions Over the Course of the Treatment
Description: Efficacy of the intake of Lpc-37 on the decrease of reported number of sleep disruptions over the course of the treatment measured with a daily online diary (mean of week summary).
  Sleep disruptions were monitored through the wash-out phase (Week 1 and 2) and the subsequent treatment phase (Weeks 3-7). In the count version, the value can be 0 or a natural number for each day and each participant. Efficacy is defined as a decrease, or (in case of a general increase) reduced increase for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group. Time is coded as a continuous variable with one value for each day and participant. Values reflect summary measures for sleep disruptions (count) for the summed counts per participant and week.
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sleep disruptions per participant & week
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
sleep disruptions per participant & week
  Week 1 (run-in) | 7.30 (6.87) | 6.09 (4.96)
  Week 2 (run-in) | 5.50 (4.62) | 5.49 (4.82)
  Week 3 (treatment) | 4.89 (5.11) | 5.11 (4.89)
  Week 4 (treatment) | 5.43 (9.20) | 4.30 (6.05)
  Week 5 (treatment) | 3.52 (3.48) | 3.53 (3.80)
  Week 6 (treatment) | 3.80 (7.40) | 4.02 (4.68)
  Week 7 (treatment) | 4.66 (6.37) | 5.83 (6.23)

27. Secondary Outcome: Change of Perceived Health Status Scores Over the Course of the Treatment
Description: Efficacy of the intake of Lpc-37 on the increase of perceived health status scores over the course of the treatment.
  Measured with a daily online diary. Health status was rated by participants on an 11-point scale (0-10; "not at all" to "very") and monitored through the wash-out phase (week 1 and 2) and the subsequent treatment phase (weeks 3-7). Higher scores indicate a high perceived health.Efficacy is defined as an increase, or (in case of a general decrease) reduced decrease for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group. Time is coded as a continuous variable with one value for each day and participant. Values reflect summary measures for perceived health status on a scale from 0 to 10 for the averaged ratings per participant and week.
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
score
  Week 1 (run-in) | 7.80 (1.31) | 7.86 (1.08)
  Week 2 (run-in) | 7.89 (1.15) | 7.92 (1.12)
  Week 3 (treatment) | 7.88 (1.20) | 7.92 (1.06)
  Week 4 (treatment) | 7.91 (1.18) | 8.01 (1.05)
  Week 5 (treatment) | 8.05 (1.22) | 7.92 (1.16)
  Week 6 (treatment) | 8.11 (1.20) | 7.73 (1.26)
  Week 7 (treatment) | 7.91 (1.15) | 7.75 (1.52)

28. Secondary Outcome: Change of Mood Scale Scores Over the Course of the Treatment
Description: Efficacy of the intake of Lpc-37 on the increase of mood scale scores over the course of the treatment
  Measured with a daily online diary. Mood was rated by participants on an 11-point scale (0-10; "very bad" to "very well") and monitored through the washout phase (week 1 and 2) and the subsequent treatment phase (weeks 3-7). Higher scores indicate a better mood. Efficacy is defined as an increase, or (in case of a general decrease) reduced decrease for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group. Time is coded as a continuous variable with one average value for each week and participant. Values reflect summary measures for mood ratings on a scale from 0 to 10 for the averaged ratings per participant and week.
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
score
  Week 1 (run-in) | 7.31 (1.25) | 7.27 (1.04)
  Week 2 (run-in) | 7.53 (1.21) | 7.49 (1.10)
  Week 3 (treatment) | 7.66 (1.05) | 7.46 (1.13)
  Week 4 (treatment) | 7.77 (1.25) | 7.53 (1.15)
  Week 5 (treatment) | 7.73 (1.17) | 7.50 (1.24)
  Week 6 (treatment) | 7.90 (1.10) | 7.40 (1.21)
  Week 7 (treatment) | 7.77 (1.30) | 7.55 (1.22)

29. Secondary Outcome: Change of Perceived Productivity Scores Over the Course of the Treatment
Description: Efficacy of the intake of Lpc-37 on the increase of perceived productivity scores over the course of the treatment
  Measured with a daily online diary. Productivity was rated by participants on an 11-point scale (0-10; "not at all" to "very") and monitored through the wash-out phase (week 1 and 2) and the subsequent treatment phase (weeks 3-7). Higher scores indicate a higher perceived productivity. Efficacy is defined as an increase, or (in case of a general decrease) reduced decrease for the active treatment group as compared to the placebo group and operationalized as the interaction between time and treatment group.Time is coded as a continuous variable with one value for each day and participant. The values reflect summary measures for perceived productivity on a scale from 0 to 10 for the averaged ratings per participant and week.
Time Frame: Daily for 2 weeks before treatment intake and 5 weeks during treatment intake
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 44 | 47
score
  Week 1 (run-in) | 6.98 (1.02) | 7.15 (1.07)
  Week 2 (run-in) | 7.34 (1.06) | 7.29 (1.03)
  Week 3 (treatment) | 7.53 (0.97) | 7.30 (1.01)
  Week 4 (treatment) | 7.48 (1.19) | 7.34 (1.18)
  Week 5 (treatment) | 7.59 (1.04) | 7.43 (1.17)
  Week 6 (treatment) | 7.57 (1.13) | 7.31 (1.22)
  Week 7 (treatment) | 7.50 (1.17) | 7.32 (1.25)

30. Secondary Outcome: The Change of the Difference From Baseline and 5 Weeks of Treatment to the Respective Mean of CAR AUCg Measures
Description: Efficacy of the intake of Lpc-37 on the reduction of the difference of Cortisol Awakening Response (CAR) area under the curve with respect to the ground (AUCg) values to the respective mean before and after 5 weeks of treatment.
  The CAR is summarized in the variables AUCg, AUCi, mean increase and peak value. These cortisol indices are frequently used to describe hypothalamic-pituitary-adrenal axis activity and represent information either of the total cortisol production or of the change in cortisol levels. AUCg is the total area under the curve of all measurements (i.e., the intensity or magnitude of the response).
  Efficacy for the CAR variables AUCg is defined in terms of a normalization: Number of participants with normal values (between first and third quantile of reference measures) and numbers of participants with low or high values are compared before treatment and after treatment. More participants in the normal range after treatment is defined as efficacy.
Time Frame: Baseline (average of 2 days before first product intake) and end of study (average of 2 days before last product intake)
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 53 | 55
number of participants
  Baseline (<25% quantile) | 6 | 12
  Baseline (25% - 75% quantile) | 36 | 30
  Baseline (>75% quantile) | 11 | 13
  End of Study (<25% quantile) | 11 | 7
  End of Study (25% - 75% quantile) | 28 | 35
  End of Study (>75% quantile) | 14 | 13

31. Secondary Outcome: The Change of the Difference From Baseline and 5 Weeks of Treatment to the Respective Mean of Cortisol Awakening Response (CAR) AUCi Measures
Description: Efficacy of the intake of Lpc-37 on the reduction of the difference of CAR area under the curve with respect to the increase (AUCi) values to the respective mean before and after the treatment.
  The CAR is summarized in the variables AUCg, AUCi, mean increase and peak value. These cortisol indices are frequently used to describe hypothalamic-pituitary-adrenal axis activity and represent information either of the total cortisol production or of the change in cortisol levels. AUCi is calculated with reference to the baseline measurement and it ignores the distance from zero for all measurements and emphasizes the changes over time. Efficacy for the CAR variables AUCi is defined in terms of a normalization: Number of participants with normal values (between first and third quantile of reference measures) and numbers of participants with low or high values are compared before treatment and after treatment. More participants in the normal range after treatment is defined as efficacy.
Time Frame: as for outcome 30
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 53 | 55
number of participants
  Baseline (<25% quantile) | 16 | 22
  Baseline (25% - 75% quantile) | 34 | 28
  Baseline (>75% quantile) | 3 | 5
  End of Study (<25% quantile) | 15 | 15
  End of Study (25% - 75% quantile) | 34 | 36
  End of Study (>75% quantile) | 4 | 4

32. Secondary Outcome: The Change of the Difference From Baseline and 5 Weeks of Treatment to the Respective Mean of Cortisol at Awakening Measures
Description: Efficacy of the intake of Lpc-37 on the reduction of the difference of Cortisol at Awakening values to the respective mean before and after 5 weeks of treatment
  Efficacy for the CAR variable cortisol at awakening is defined in terms of a normalization: Number of participants with normal values (between first and third quantile of reference measures) and numbers of participants with low or high values are compared before treatment and after treatment. More participants in the normal range after treatment is defined as efficacy.
Time Frame: as for outcome 30
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 53 | 55
number of participants
  Baseline (<25% quantile) | 14 | 16
  Baseline (25% - 75% quantile) | 31 | 26
  Baseline (>75% quantile) | 8 | 13
  End of Study (<25% quantile) | 19 | 12
  End of Study (25% - 75% quantile) | 26 | 34
  End of Study (>75% quantile) | 8 | 9

33. Secondary Outcome: The Change of the Difference From Baseline and 5 Weeks of Treatment to the Respective Mean of CAR 8pm Measures
Description: Efficacy of the intake of Lpc-37 on the reduction of the difference of cortisol at 8 pm values to the respective mean before and after 5 weeks of treatment
  Efficacy for the CAR variable cortisol at 8 pm is defined in terms of a normalization: Number of participants with normal values (between first and third quantile of reference measures) and numbers of participants with low or high values are compared before treatment and after treatment. More participants in the normal range after treatment is defined as efficacy.
Time Frame: Baseline (average of 2 days before first product intake) and end of study (average of 2 days before last product intake
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | Lpc-37 | Placebo
Number analyzed (Participants) | 53 | 55
number of participants
  Baseline (<25% quantile) | 4 | 6
  Baseline (25% - 75% quantile) | 20 | 23
  Baseline (>75% quantile) | 29 | 26
  End of Study (<25% quantile) | 3 | 7
  End of Study (25% - 75% quantile) | 28 | 18
  End of Study (>75% quantile) | 22 | 30

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected daily during the 5-week intervention period and tracked when the AE continued at the end of the study (up to 30 days afterwards)
Description: AE reporting was done by the Investigator or her designees. All AEs were collected on the paper case report forms.
  Variables recorded for each AE: Description of the event, onset and resolution (date and time), whether the AE is ongoing at the end of the study, intensity (mild, moderate, severe), therapy of event, action taken, outcome, causality (definitely, probably, possibly, unlikely, not related, not assessable) and whether it constitutes an Serious Adverse Event (SAE) or not.
Arm/Group | Lpc-37 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 29/59 | 26/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lpc-37 (N=59) | Placebo (N=59)
common cold (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 4 (4)
sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 8 (10)
headache (Nervous system disorders) | 22 (34) | 15 (34)
stomach ache (Gastrointestinal disorders) | 5 (8) | 7 (10)
Head cold (Infections and infestations) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Vertigo (Cardiac disorders) | 2 (2) | 4 (4)
Discomfort/Complaints related to the menstrual cycle (General disorders) | 2 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Overall Non-disclosure and Confidentiality Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT03494725/Prot_SAP_000.pdf